CLINICAL TRIAL: NCT07117708
Title: The Optimize Trial: Optimizing Timing of Cesarean Delivery Consent on Labor and Delivery
Brief Title: Optimizing Timing of Cesarean Delivery Consent on Labor and Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00117303
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; Informed Consent
Keywords: pregnancy; informed consent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Consent for Possible Cesarean Delivery (Experimental): Patients randomized to this arm of the study will undergo surgical consent for possible cesarean delivery upon arrival to labor and delivery for the start of their induction of labor.
  Interventions: Other: Early Surgical Consent
- Indicated Consent for Possible Cesarean Delivery (Active Comparator): Patients randomized to this arm of the study will undergo surgical consent for possible cesarean delivery only if it appears to be clinically indicated throughout their induction of labor.
  Interventions: Other: Surgical Consent if Clinically Indicated

INTERVENTIONS:
Other: Early Surgical Consent — Surgical consent for possible cesarean delivery will be completed upon arrival to labor and delivery before induction of labor begins
  Arms: Early Consent for Possible Cesarean Delivery
Other: Surgical Consent if Clinically Indicated — Surgical consent for possible cesarean delivery will be completed if it appears clinically indicated during a participant's induction of labor.
  Arms: Indicated Consent for Possible Cesarean Delivery

SUMMARY:
Nationally, 32.1% of pregnant patients deliver via cesarean delivery, including both patients who undergo a planned cesarean delivery and patients who intend to undergo vaginal delivery and are recommended to deliver via cesarean delivery. The investigators aim to understand how to optimize the patient experience for patients who present to the hospital intending to deliver vaginally but are recommended to deliver via cesarean delivery (an unplanned cesarean delivery). Practices regarding timing of informed consent for possible cesarean delivery vary widely across hospitals in the United States; some institutions will consent every patient on admission to the hospital for possible cesarean delivery, whereas some institutions consent patients for possible cesarean delivery only if a patient's clinical course suggests cesarean delivery may be indicated.

This study aims to determine optimal timing for consent for possible cesarean delivery by randomizing patients to either be consented for possible cesarean delivery on admission to the hospital or if it appears to be clinically indicated. This study will only assess altered timing of a surgical consent process and will not impact the clinical care participants receive. After delivery, participants will share their experiences with the consent process and with their overall childbirth experience.

DETAILED DESCRIPTION:
This study is a randomized-controlled trial in which patients presenting to Labor and Delivery for their scheduled induction of labor will be randomized to either be consented for possible cesarean delivery on admission to Labor and Delivery or be consented for possible cesarean delivery if it appears to be clinically indicated (as is current standard of care). The purpose of this study is to understand whether earlier cesarean delivery consent could be one strategy to improve the delivery experience of patients recommended to undergo unplanned cesarean delivery and enhance education for all birthing patients. The proposed study will fill this gap in the literature by determining whether early informed surgical consent reduces negative patient delivery experiences and address concerns about the mechanism of obtaining informed consent for cesarean delivery.

Duke Perinatal Durham or Duke Women's Health Associates patients will be approached to be consented for the research study between 34-41 weeks of pregnancy. Those who agree to participate will be randomized to either an early surgical consent for possible cesarean delivery at the time of admission to Labor and Delivery or, as per our current standard of care, will be surgically consented for cesarean delivery if it is clinically indicated. On postpartum day 1, patients will be texted a link to a survey about their experience with the surgical consent process and their overall childbirth experience. The investigators will collect additional patient information via chart review, including a patient's medical history and information about their labor, delivery, and postpartum courses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Receiving prenatal care at Duke Perinatal Durham or Duke Women's Health Associates
* Between 34 weeks 0 days and 41 weeks 0 days of gestation
* Scheduled for induction of labor OR are eligible/intend to be scheduled for an induction of labor

Exclusion Criteria:

* Trial of labor after cesarean delivery
* Multiple gestation
* Major fetal anomalies
* Presenting for induction of labor as a transfer from the antepartum inpatient service
* Non-English speaking
* Those who do not intend to labor
* Patients who are ineligible for vaginal delivery for other reasons, including fetal malpresentation or abnormal placentation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Patient Perception of Informed Consent Process | From day 1 postpartum to 6 weeks postpartum
  As measured by survey.

SECONDARY OUTCOMES:
Patient Childbirth Experience | From day 1 postpartum to 6 weeks postpartum
  As measured by survey.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Beal, Study Director — Duke University Department of Obstetrics and Gynecology; Kristin Weaver, Study Director — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burcher P, Hushmendy S, Chan-Mahon M, Dasani M, Gabriel J, Crosby E. Unplanned Cesarean Birth: Can the Quality of Consent Affect Birth Experiences? AJOB Empir Bioeth. 2020 Oct-Dec;11(4):268-274. doi: 10.1080/23294515.2020.1817174. Epub 2020 Sep 18. PMID 32945733
- [Background] Fink AS, Prochazka AV, Henderson WG, Bartenfeld D, Nyirenda C, Webb A, Berger DH, Itani K, Whitehill T, Edwards J, Wilson M, Karsonovich C, Parmelee P. Predictors of comprehension during surgical informed consent. J Am Coll Surg. 2010 Jun;210(6):919-26. doi: 10.1016/j.jamcollsurg.2010.02.049. PMID 20510800
- [Background] Salmeen K, Brincat C. Time from consent to cesarean delivery during labor. Am J Obstet Gynecol. 2013 Sep;209(3):212.e1-6. doi: 10.1016/j.ajog.2013.05.004. Epub 2013 May 6. PMID 23659991
- [Background] Odumosu M, Pathak S, Barnet-Lamb E, Akin-Deko O, Joshi V, Selo-Ojeme D. Understanding and recollection of the risks associated with cesarean delivery during the consent process. Int J Gynaecol Obstet. 2012 Aug;118(2):153-5. doi: 10.1016/j.ijgo.2012.03.025. Epub 2012 May 1. PMID 22554992
- [Background] Akkad A, Jackson C, Kenyon S, Dixon-Woods M, Taub N, Habiba M. Informed consent for elective and emergency surgery: questionnaire study. BJOG. 2004 Oct;111(10):1133-8. doi: 10.1111/j.1471-0528.2004.00240.x. PMID 15383117
- [Background] Lescale KB, Inglis SR, Eddleman KA, Peeper EQ, Chervenak FA, McCullough LB. Conflicts between physicians and patients in non-elective cesarean delivery: incidence and the adequacy of informed consent. Am J Perinatol. 1996 Apr;13(3):171-6. doi: 10.1055/s-2007-994319. PMID 8688110
- [Background] Levy KS, Smith MK, Lacroix M, Yudin MH. Patient Satisfaction with Informed Consent for Cesarean and Operative Vaginal Delivery. J Obstet Gynaecol Can. 2022 Jul;44(7):785-790. doi: 10.1016/j.jogc.2022.03.010. Epub 2022 Mar 29. PMID 35364294
- [Background] Ryding EL, Wijma B, Wijma K. Posttraumatic stress reactions after emergency cesarean section. Acta Obstet Gynecol Scand. 1997 Oct;76(9):856-61. doi: 10.3109/00016349709024365. PMID 9351412
- [Background] Olde E, van der Hart O, Kleber R, van Son M. Posttraumatic stress following childbirth: a review. Clin Psychol Rev. 2006 Jan;26(1):1-16. doi: 10.1016/j.cpr.2005.07.002. Epub 2005 Sep 19. PMID 16176853
- [Background] Blomquist JL, Quiroz LH, Macmillan D, McCullough A, Handa VL. Mothers' satisfaction with planned vaginal and planned cesarean birth. Am J Perinatol. 2011 May;28(5):383-8. doi: 10.1055/s-0031-1274508. Epub 2011 Mar 4. PMID 21380993
- [Background] Smarandache A, Kim TH, Bohr Y, Tamim H. Predictors of a negative labour and birth experience based on a national survey of Canadian women. BMC Pregnancy Childbirth. 2016 May 18;16(1):114. doi: 10.1186/s12884-016-0903-2. PMID 27193995
- [Background] Osterman MJK, Hamilton BE, Martin JA, Driscoll AK, Valenzuela CP. Births: Final Data for 2022. Natl Vital Stat Rep. 2024 Apr;73(2):1-56. PMID 38625869